CLINICAL TRIAL: NCT01144884
Title: Development of a Clinical Prediction Rule to Identify Patients With Neck Pain Likely to Benefit From Education and Exercise
Brief Title: Identify Patients With Neck Pain Likely to Benefit From Education and Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William J. Hanney (Other)
Collaborators: Nova Southeastern University (Other); Franklin Pierce University (Other); AdventHealth (Other)
Responsible Party: Sponsor-Investigator, William J. Hanney, Assistant Professor, University of Central Florida
Organization: University of Central Florida (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18808040
Record Dates: First submitted 2010-06-09; First posted 2010-06-16 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Neck Pain
Keywords: Neck pain; education; exercise; clinical prediction rule
MeSH Terms: conditions — Neck Pain; Motor Activity | interventions — Educational Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm trial (Other): Education:To standardize, treatment education will consist of counsel to stay active. Details will be given to subjects verbally & reinforced in the home booklet.
  Posture:Facilitation of proper posture has been show to increase recruitment of the lumbar multifidus & deep neck flexors. Instruction will be given verbally & in writing.
  Stretching:Stretching exercises will be targeted to address these common impairments. Patients will be introduced to proper stretching procedures. Each stretch will be held for 30s & repeated two times,each side as applicable. The following stretches will be performed:
  Upper trap Anterior/medial Scalene Suboccipital Pectoralis
  Muscular Performance: Muscle performance will be trained incorporating components of strength, endurance and motor control. Each of the exercises listed below are outlined based on progressions.
  Isometric Cervical Extension Craniocervical flexion Seated Row Seated "T" Palms Up Seated Side Arm Raises
  Interventions: Other: Procedure (education and exercise)

INTERVENTIONS:
Other: Procedure (education and exercise) — education/exercise

SUMMARY:
The annual incidence of neck pain has been reported to be 14.6%. Other studies outline a wide disparity in the lifetime incidence of neck pain ranging from 22% to 70%. Numerous treatment options exist for the management of neck pain however, there is limited evidence to support which interventions are most effective. Exercise based interventions are commonly used in the treatment of patients with neck pain however; it is not clear which patients are most likely to benefit from this type of treatment. The purpose of this project is to develop a clinical prediction rule (CPR) to identify which patients with neck pain have a greater probability of benefiting from a standardized program of education and exercise. Ninety (90) patients referred to physical therapy will undergo a standardized examination to assess potential predictor variables. Upon completion of the examination a standardized treatment program of education and exercise will be administered regardless of examination findings. Self report measures will be administered on the initial examination and on follow up visits at 2, 4, and 6 weeks. A questionnaire and outcome measures will be also mailed out 6 months after initiation of treatment to assess long-term change. Once the treatment plan is completed, patients will be classified as having either a successful or non-successful response. Subjects which rated their perceived recovery on the Global Rating of Chance (GROC) as "a very great deal better", "a great deal better", "quite a bit better", or "moderately better" (i.e., a score of +4 or greater) will be categorized as having a successful outcome. The primary endpoints to determine the outcome will be analyzed at 6 weeks and 6 months. The result of this study will assist physical therapists to identify sub-groups of patients likely to benefit from a program of education and exercise. The categorization of patients in groups based on beneficial treatments may help to provide improved outcomes.

DETAILED DESCRIPTION:
The sample size will consist of 90 subjects ages 18 or above with a primary complaint of neck pain. The subjects must be able to read and communicate in English in order to complete the required documentation. No specific conditions are to be included which would make this a protected population.

Patients will be recruited in one of two ways. First, flyers will be sent to local referrals announcing the study and request for subjects. Should a patient be interested in participating they will call the PI at the phone number listed on the flyer. The PI will inquire about patient location and coordinate a convenient location. Second, patients which present to a participating clinic with primary complaint of neck pain will be handed a flyer and asked by the front office if they would be interested to hear more about the study. If the patient expresses interest in participating they will meet with a clinician trained in the study to review inclusion and exclusion criterion. Should the patient meet all inclusion and have no exclusion criterion, the informed consent form will be reviewed with the patient by a trained clinician. Once the patient has agreed to participate and signed the informed consent they will be formally enrolled into the study.

All information obtained in this study is strictly confidential unless disclosure is required by law. Federal Privacy Regulations provide safeguards for privacy, security, and authorized access. Except when required by law, the patient will not be identified by name, social security number, address, telephone number, or any other direct personal identifier.

All records pertaining to the patient's involvement in this research study will be stored in a locked file cabinet. A case number will indicate the patient's identity on these records. This information will only be accessible to the investigators listed on the first page of this document and the research study staff.

Methods and Procedures This study will follow a standardized examination and treatment protocol. All interventions and techniques have been proven to be effective in this patient population. Once the patient is deemed eligible for the study the informed consent will be reviewed by an investigator. If the patient agrees to participate in the study they will sign the informed consent. The patient will complete self report measures which will take approximately 20 minutes. Self report measures to be completed include the neck disability index (NDI), fear avoidance beliefs questionnaire (FABQ), global rating of change (GROC), and numeric pain rating scale (NPRS). An investigator will then perform a standardized examination which will take approximately 1 hour. Examination findings will be recorded on the cervical examination form. The patient will then be given an opportunity to undergo a second examination by a blinded examiner for reliability purposes. This second examination is optional and must be performed within 48 hours and before treatment is initiated.

Upon completion of the examination the patient will be issued a home care guide which included educational materials and the standardized exercise program. The patients will be asked to review the educational information. When the patient returns for follow up visits the standardized treatment program of education and exercise will be initiated and progressed. Each subsequent treatment session will last approximately one hour. The patient will be asked to perform the exercise program 2 times per week for 6 weeks and perform stretches independently. In order to monitor progress the self report measures will be completed every two weeks.

When applicable, a portion of the research costs associated with the physical therapy procedures will be billed to the patient's insurance provider. The patient's co-payments will be the same as if they were not part of the research study. The procedures will be documented in their medical/Research record. There will be no additional costs to the patient outside of the normal delivery of care and no further payment will be offered to the patient for participation in the study. Participants will be reimbursed a nominal amount for the time necessary to complete the research documentation. Subject reimbursement is as follows:

Data Analysis Reliability of the examination variables will be assessed for a blinded examiner on a second examination. Descriptive statistics will be calculated which include frequency counts for categorical data and calculation of the mean and standard deviation (SD) for continuous variables. Cohen k will be used to calculate inter-rater reliability of categorical data with only 2 response options possible. A weighted k will be used to calculate the reliability of categorical data with 3 response options. The weight k will be calculated using a linear weighting method. Intraclass correlation coefficients (ICC) model 2,1 and the 95% confidence intervals will be calculated to determine the inter-rater reliability for continuous variables. The standard error of measurement (SEM) will be calculated as SD√ (1-r), where SD is the standard deviation of the observed scores and r is the reliability coefficient for the measurement. The minimal detectable change (MDC) for continuous variables will be calculated as 1.96X SEM X √2. The total measure of error will be calculated for continuous data by mean difference between raters (rater A - rater B) +/- 1.96 X SD. The total measure of error represents the values within which 95% of the measurements between raters lie. Reliability for categorical variables will be interpreted as follows; values < 0.10 no agreement; 0.11 to 0.40 slight agreement; 0.41 to 0.60 fair agreement; 0.61 and 0.80 moderate agreement and values >0.81 substantial agreement. Reliability for continuous variables will be interpreted as follows: < 0.10 no agreement; 0.11 to 0.40 slight agreement; 0.61 and 0.80 moderate agreement; and values > 0.81 substantial agreement.

Dependent t-tests will be used to analyze each of the primary outcome variables including Numeric pain rating scale (NPRS), Neck Disability Index (NDI), Fear Avoidance Beliefs Questionnaire - Physical Activity (FABQ-PA) and Fear Avoidance Beliefs Questionnaire - Work (FABQ-W). The alpha level will be set at 0.05. Multiple comparisons will be conducted (baseline - 2 weeks; baseline - 4 weeks; baseline - 6 weeks and baseline - 6 months) between the paired time frames with a dependent t-test. Bonferroni correction will be used to establish the significance level at 0.0125 (.05/4).

Potential predictor variables will come from the outcome measures, demographics form, history and physical assessment. Analysis will be implemented using independent t-tests for continuous variables and X2 tests for categorical variables to determine differences between successful and non-success outcomes. Variables with a significance of p<.10 will be retained as potential prediction variables for each group. This p value will be used to decrease the likelihood that a potential predictor variable will be missed. Sensitivity and specificity values will be calculated for continuous variables with a significant univariate relationship and plotted as a receiver operating characteristics (ROC) curve. The point on the curve which is closest to the upper left corner represents the values with greatest diagnostic accuracy. This point will be selected as the cutoff defining a positive test. Sensitivity, specificity and likelihood ratios will be calculated for retained variables in the successful and non-successful groups. Potential predictor variables for each group will then be entered into a separate backward stepwise logistic regression model to identify the most prudent group of variables for the treatment outcome. Those variables preserved in the regression model will be used to develop a multivariate CPR for classifying patients likely to have a successful and non-successful outcome by completing a program of education and exercise for this sample.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18
2. Primary complaint of neck pain with or without unilateral UE symptoms
3. Neck Disability Index (NDI) of 10% or greater.

Exclusion Criteria:

1. Presence of medical "red flags' noted in the Neck Medical Screening Questionnaire. (i.e. tumor, fracture, etc.)
2. Evidence of central nervous system (CNS) involvement (i.e. hyperreflexia, sensory disturbances in the hand, intrinsic muscle wasting of the hands, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes such as Hoffman's or Babinski reflexes, etc.)
3. Spasmodic torticollis
4. Frequent migraine
5. Fibromyalgia
6. Prior Surgery to the neck or thoracic spine
7. Severe psychiatric illness
8. Inability to comply with treatment and follow-up schedule
9. Pending legal action regarding their neck pain
10. Insufficient English language skills to complete all questionnaires.
11. Latex allergies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2009-08; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Perceived Disability as measured by the Neck Disability Index | 6 weeks
Perceived pain intensity as measure by the Numeric pain rating scale | Baseline, 2 weeks, 4 weeks, 6 weeks, 6 months
Perceived fear avoidance beliefs as measure by the Fear Avoidance Belief Questionnaire | 6 weeks
Perceived rating of change as measure by the Global Rating of Change | 6 weeks

SECONDARY OUTCOMES:
Disability as measured by the Neck Disability Index | baseline, 2 weeks, 4 weeks, 6 months
Perceived pain intensity as measure by the Numeric pain rating scale | baseline, 2 weeks, 4 weeks, 6 months
Perceived fear avoidance beliefs as measure by the Fear Avoidance Belief Questionnaire | baseline, 2 weeks, 4 weeks, 6 months
Perceived rating of change as measure by the Global Rating of Change | 2 weeks, 4 weeks, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: William Hanney, PT DPT, Principal Investigator — University of Central Florida
Locations (9):
- United States (9):
  - Florida Hospital Sports Medicine & Rehabilitation - Altamonte, Altamonte Springs, Florida
  - Brooks Rehabilitation - Monument, Jacksonville, Florida
  - Brooks Rehabilitation -Spine Center, Jacksonville, Florida
  - Florida Hospital Sports Medicine & Rehabilitation - Kissimmee, Kissimmee, Florida
  - Brooks Rehabilitation - Lake Mary, Lake Mary, Florida
  - Brooks Rehabilitation - Flemming Island, Orange Park, Florida
  - Florida Hospital Sports Medicine & Rehabilitation - RDV, Orlando, Florida
  - Brooks Rehabilitation - Waterford, Orlando, Florida
  - Florida Hospital Sports Medicine & Rehabilitation - Oviedo, Oviedo, Florida